CLINICAL TRIAL: NCT06315153
Title: Research of Comprehensive Assessment of Carotid Plaque Vulnerability and Development of Atherosclerotic Ischemic Stroke Risk Prediction Model
Brief Title: Comprehensive Assessment of Atherosclerotic Ischemic Stroke Risk and Development of a Prediction Model
Acronym: CAIS-pre
Status: Active, not recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: KS2023077-1
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-05

CONDITIONS: Carotid Stenosis; Ischemic Stroke
Keywords: plaque vulnerability; vascular ultrasound; atherosclerosis; ischemic stroke; contrast-enhanced ultrasound
MeSH Terms: conditions — Carotid Stenosis; Ischemic Stroke; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — This study does not involve specimen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- symptomatic group: An ischemic stroke was defined as occurring if the patient developed clinical symptoms related to neurological deficits and/or new infarcted lesions were detected on magnetic resonance imaging, and patients who developed ischemic strokes were classified in the symptomatic group.
- asymptomatic group: Patients without an ischemic stroke were classified in the asymptomatic group.

SUMMARY:
This observational study was designed for the assessment of plaque vulnerability in patients with carotid atherosclerotic stenosis and the development of predictive models for the occurrence and recurrence of atherosclerotic ischemic stroke.

The objectives of the study were as follows: first, to integrate the degree of carotid stenosis and plaque characteristics assessed by vascular ultrasound for a comprehensive assessment of plaque vulnerability; second, to develop an assessment tool for the risk of future ischemic stroke in patients with asymptomatic carotid stenosis by combining vascular risk factors, serologic markers, carotid ultrasound characteristics, and contrast-enhanced ultrasonographic parameters; and third, to incorporate vascular ultrasound parameters into existing predictive models of ischemic stroke recurrence risk to develop a risk assessment tool for atherosclerotic ischemic stroke.

The main questions it aims to answer are:

* How to screen high-risk patients and those eligible for revascularization from asymptomatic carotid stenosis patients for primary prevention of stroke.
* How to improve the prediction accuracy of atherosclerotic ischemic stroke based on existing prediction models for secondary prevention of stroke.

DETAILED DESCRIPTION:
The data from January 2022 to December 2022 was obtained from the electronic medical record system, but there will be a two-year follow-up of the data. Therefore, this is a two-way cohort study, containing both a retrospective and prospective cohort.

ELIGIBILITY:
Inclusion Criteria:

* ① Patients aged ≥ 40 years old; ② Complete clinical data and serological indicators; ③ Carotid artery ultrasound examination was performed after admission.

Exclusion Criteria:

* ① Unilateral or bilateral carotid artery occlusion; ②Carotid stenosis caused by other reasons, such as entrapment, aortitis, radiculopathy and muscle fiber dysplasia; ③Previous carotid stenting or carotid endarterectomy; ④Carotid artery plaques are strongly echogenic with acoustic shadowing, resulting in unclear detection of the lumen.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Five hundred hospitalized patients with ≥50% carotid artery stenosis between January 2022 and January 2024 were collected, including 400 in Xuanwu Hospital of Capital Medical University and 100 in the First Hospital of Jilin University.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
The occurrence of ischemic stroke | 2 years
  Clinical symptoms related to neurological deficits in patients and/or discovery of new infarcted lesions on head magnetic resonance imaging/computed tomography scans
The recurrence of ischemic stroke | 2 years
  Clinical symptoms related to neurological deficits in patients and/or discovery of new infarcted lesions on head magnetic resonance imaging/computed tomography scans

CONTACTS AND LOCATIONS:
Overall Officials: Yingqi Xing, PhD, Study Chair — Xuanwu Hospital, Beijing
Locations (2):
- China (2):
  - The first hospital of Jilin university, Changchun, Jilin
  - Xuanwu Hospital, Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaudhary D, Abedi V, Li J, Schirmer CM, Griessenauer CJ, Zand R. Clinical Risk Score for Predicting Recurrence Following a Cerebral Ischemic Event. Front Neurol. 2019 Nov 12;10:1106. doi: 10.3389/fneur.2019.01106. eCollection 2019. PMID 31781015
- [Background] Fedak A, Ciuk K, Urbanik A. Ultrasonography of vulnerable atherosclerotic plaque in the carotid arteries: B-mode imaging. J Ultrason. 2020;20(81):e135-e145. doi: 10.15557/JoU.2020.0022. Epub 2020 Jun 15. PMID 32609972
- [Background] Saba L, Saam T, Jager HR, Yuan C, Hatsukami TS, Saloner D, Wasserman BA, Bonati LH, Wintermark M. Imaging biomarkers of vulnerable carotid plaques for stroke risk prediction and their potential clinical implications. Lancet Neurol. 2019 Jun;18(6):559-572. doi: 10.1016/S1474-4422(19)30035-3. Epub 2019 Apr 4. PMID 30954372
- [Background] van Dam-Nolen DHK, Truijman MTB, van der Kolk AG, Liem MI, Schreuder FHBM, Boersma E, Daemen MJAP, Mess WH, van Oostenbrugge RJ, van der Steen AFW, Bos D, Koudstaal PJ, Nederkoorn PJ, Hendrikse J, van der Lugt A, Kooi ME; PARISK Study Group. Carotid Plaque Characteristics Predict Recurrent Ischemic Stroke and TIA: The PARISK (Plaque At RISK) Study. JACC Cardiovasc Imaging. 2022 Oct;15(10):1715-1726. doi: 10.1016/j.jcmg.2022.04.003. Epub 2022 Jun 15. PMID 36202450